CLINICAL TRIAL: NCT04670055
Title: Clinical Trial for the Safety and Efficacy of Humanized BCMA-targeted CAR-T Cells Therapy for Refractory/Relapsed Multiple Myeloma
Brief Title: A Study of Humanized BCMA-targeted CAR-T Cells Therapy for Refractory/Relapsed Multiple Myeloma
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Yake Biotechnology Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, Clinical Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: hBCMA-ZhejiangU
Record Dates: First submitted 2020-12-09; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Relapse Multiple Myeloma; Refractory Multiple Myeloma
Keywords: multiple myeloma; CAR T-cell therapy; BCMA
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Administration of BCMA Targeted CAR T-cells (Experimental): Dose escalation follows the standard 3+3 dose escalation design. A total of 3 dose levels are set for subjects.
  Interventions: Drug: BCMA Targeted CAR T-cells

INTERVENTIONS:
Drug: BCMA Targeted CAR T-cells — Each subject receive BCMA Targeted CAR T-cells by intravenous infusion
  Other Names: BCMA Targeted CAR T-cells injection

SUMMARY:
Clinical Trial for the safety and efficacy of humanized BCMA-targeted CAR-T cells therapy for refractory/relapsed multiple myeloma

DETAILED DESCRIPTION:
This is a single arm, open-label, single-center study. This study is indicated for relapsed BCMA+ multiple myeloma, the selections of dose levels and the number of subjects are based on clinical trials of similar foreign products. 50 patients will be enrolled for this trial. Primary objective is to explore the safety, main consideration is dose-related safety.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of multiple myeloma (MM):

   1. Patients with BCMA positive relapsed/refractory MM;
   2. Relapsed after hematopoietic stem cell transplantation;
   3. Cases with recurrent positive minimal residual disease;
   4. Extramedullary leision which is hard to be eradicated by chemotherapy or radiotherapy.
2. Anticipated survival time more than 12 weeks;
3. Male or female aged 30-75 years;
4. Those who voluntarily participated in this trial and provided informed consent.

Exclusion Criteria:

Subjects with any of the following exclusion criteria were not eligible for this trial:

1. History of craniocerebral trauma, conscious disturbance, epilepsy, cerebrovascular ischemia, and cerebrovascular hemorrhagic diseases;
2. Electrocardiogram shows prolonged QT interval, severe heart diseases such as severe arrhythmia in the past;
3. Pregnant (or lactating) women;
4. Patients with severe active infections (excluding simple urinary tract infection and bacterial pharyngitis);
5. Active infection of hepatitis B virus or hepatitis C virus;
6. Concurrent therapy with systemic steroids within 2 weeks prior to screening, except for the patients recently or currently receiving in haled steroids;
7. Previously treated with any CAR-T cell product or other genetically-modified T cell therapies;
8. Creatinine>2.5mg/dl, or ALT / AST > 3 times of normal amounts, or bilirubin>2.0 mg/dl;
9. Other uncontrolled diseases that were not suitable for this trial;
10. Patients with HIV infection;
11. Any situations that the investigator believes may increase the risk of patients or interfere with the results of study.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Baseline up to 28 days after BCMA targeted CAR T-cells infusion
  Adverse events assessed according to NCI-CTCAE v5.0 criteria
Incidence of treatment-emergent adverse events (TEAEs) | Up to 2 years after BCMA targeted CAR T-cells infusion
  Incidence of treatment-emergent adverse events [Safety and Tolerability]

SECONDARY OUTCOMES:
Overall response rate (ORR) | At Day 28
  Assessment of ORR at Day 28
Overall survival (OS) | At Month 6, 12, 24
  Assessment of OS at Month 6, 12, 24
Quality of life(EORTC QLQ-C30) Core 30 (EORTC QLQ-C30) | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment using European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) scale [For item1-28: max score: 112, min score: 28, higher scores mean a better outcome; for item 28-29: max score: 14, min score: 2, higher scores mean a worse outcome] to measure Quality of life at Baseline, Month 1, 3, 6, 9 and 12
Instrumental Activities of Daily Living (IADL) score | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment of Instrumental Activities of Daily Living (IADL) scale [max score: 56, min score: 14, higher scores mean a worse outcome] at Baseline, Month 1, 3, 6, 9 and 12
Activities of Daily Living (ADL) score | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment using Activities of Daily Living (ADL) scale (Barthel Index) [max score: 100, min score: 0, higher scores mean a better outcome] at Baseline, Month 1, 3, 6, 9 and 12
Hospital Anxiety and Depression Scale (HADS) score | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment of Hospital Anxiety and Depression Scale (HADS) score at Baseline, Month 1, 3, 6, 9 and 12

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Medical College, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen R, Jin C, Liu K, Zhao M, Yang T, Zhang M, Xiao P, Feng J, Hong R, Fu S, Cui J, Huang S, Wei G, Huang H, Hu Y. Predictive value of pre-treatment circulating tumor DNA genomic landscape in patients with relapsed/refractory multiple myeloma undergoing anti-BCMA CAR-T therapy: Insights from tumor cells and T cells. Chin Med J (Engl). 2024 Nov 6;138(19):2481-90. doi: 10.1097/CM9.0000000000003306. Online ahead of print. PMID 39501801